CLINICAL TRIAL: NCT01552954
Title: Effects of Low Sodium Intake on the Anti-proteinuric Efficacy of Olmesartan in Hypertensive Patients With Albuminuria Through Open-label Randomized Trial
Brief Title: Effects of Low Sodium Intake on the Anti-proteinuric Efficacy in Hypertensive Patient With Olmesartan
Acronym: ESPECIAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Daiichi Sankyo (Industry); Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Principal Investigator, Ho Jun Chin, Associate Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1112/142-008
Record Dates: First submitted 2012-02-24; First posted 2012-03-13 (Estimated); Results first posted 2014-12-18 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Hypertension; Chronic Kidney Disease; Microalbuminuria
Keywords: hypertension; Chronic kidney disease; albuminuria; low salt diet; Angiotensin II receptor blocker
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic; Albuminuria | interventions — Diet, Sodium-Restricted; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive education of low salt diet (Experimental): For 8 weeks, dietitian will call patients to take the information according to pre-defined questionnaire, to check the daily diet habit and daily food taken, and to guide how to lessen sodium intake for 30 min at each call. The call will be done once a week for 8 weeks. (*Intervention in this trial is the "intensity of education")
  Interventions: Behavioral: Intensive education of low salt diet
- Conventional diet group (No Intervention): Education for low salt diet will be conducted as in office with brief communication with a patient and a physician.

INTERVENTIONS:
Behavioral: Intensive education of low salt diet — For 8 weeks, dietitian will call patients to take the information according to pre-defined questionnaire, to check the daily diet habit and daily food taken, and to guide how to lessen sodium intake for 30 min at each call. The call will be done once a week for 8 weeks.
  Other Names: low salt diet; Angiotensin II converting enzyme; albuminuria; chronic kidney disease
  Arms: Intensive education of low salt diet

SUMMARY:
Purpose of this study

1. Intensive education for low salt diet will be enhance the anti-proteinuric effect of Olmesartan, a popular anti-hypertensive drug of angiotensin II receptor blocker, in Koreans compared to conventional prescription of medication.
2. Intensive education for low salt diet will decrease the amount of 24 hour-urine sodium excretion compared to control group, effectively.

DETAILED DESCRIPTION:
1. Background

   A. The chronic kidney disease (CKD) is the one of the main burden of chronic diseases and the prevalence of CKD is increasing in worldwide. In Korea, the prevalence of CKD was reported as 13.7% among urban Korean adults in 2008 by our study group.

   B. It is well known the CKD is the most important risk factor to cardiovascular events, cardiovascular mortality, all cause-mortality, and hospitalization. The cost of the management for the CKD was high and it took 3.25% of all budgets for medical reimbursement in 2004 for all Koreans, which was ranked on the top of expenditure for single disease category.

   C. The most popular risk factors to CKD progression are aging, obesity, hyperlipidemia, diabetes mellitus, hypertension, and proteinuria. The hypertension and proteinuria also cause the cardiovascular events and increase the mortality rate.

   D. The inhibitors for renin-angiotensin aldosterone system, angiotensin II type I receptor blocker (ARB) and angiotensin converting enzyme inhibitor (ACEI), are well known medications to prevent cardiovascular events and renal functional deterioration to end stage renal disease(ESRD) in patients with hypertension, non-diabetic CKD, or diabetic nephropathy. One of the adverse events of ARB is the decrease of hemoglobin. Inoue et al reported the level of hemoglobin was decreased in amount of 0.45 ±0.89 g/dL after prescription of ARB and valsartan decreased the erythropoietin in 6 days after medication. The exact mechanism of decrease of hemoglobin by ARB was not fully verified but it is related to decrease effects of angiotensin II on aggravating hypoxia in the kidney and on the activation of hypoxia-inducible factor 1α (HIF1a) and then decrease the production of erythropoietin as in the report of Durmus et al. Considering that the relationships between ARB usage and decrease of proteinuria in transplanted kidney, between aggravation of hypoxia or HIF1a and CKD, and between ARB and the decrease of HIF1a or erythropoietin(EPO), we could postulate that the decrease of hemoglobin would not be a adverse effect of ARB to deteriorate patients' condition but a co-phenomenon of ARB's anti-RAS effect and a marker of ARB's effectiveness.

   E. The anti-proteinuric effect of ARB is decreased by high salt intake. For example, ARB treatment without low salt intake decreased proteinuria by 30% in patients with proteinuria 2-10g/day compared to baseline value and addition of low salt diet to ARB treatment further decreased proteinuria up to 25%. But, using slow salt tablets, increase of daily intake of sodium diminished the anti-proteinuric effect of ARB in diabetic nephropathy.

   F. The previous studies for the effect of ARB on proteinuria affected by sodium intake took the methods of controlled diet by researcher or using slow salt tablet but these method are not practical to adopt in real clinical practice.

   G. The moderate and mild decrease of daily sodium intake which lower the daily excretion of sodium by 55 mEq/day had an effect of decrease of proteinuria by 11% in hypertensive patients.

   H. The mean amount of sodium of Korean diets was reported as high as 208 mmol/day in Intersalt study, which is more than 11 g of salt. The recent reports also showed the trend of high salt-intake by Koreans.
2. Rationale So, It is worth to do this study because

   * high salt intake is prevalent in Koreans,
   * high salt diet diminishes the effect of ARB on proteinuria
   * the methods used in previous studies were not suitable to apply to clinical practice,
   * and there were no study to reveal the decrease of hemoglobin would the marker for the effect of ARB and not be a adverse event of ARB.
3. Objectives

   1. Primary objective: The difference between amount of albuminuria after usage of Olmesartan and amount of albuminuria after prescription of Olmesartan with intensive diet education in intervention group is higher than the difference of albuminuria in control group.
   2. Secondary objective:

   Item 1: In all patients, Olmesartan decreases the albuminuria. Item 2: In all patients, the change of hemoglobin after prescription of Olmesartan is proportional to the change of albuminuria and serum erythropoietin.

   Item 3: Intensive education for low salt diet induces the significant decrease of daily sodium excretion in Intervention group compared to control group.

   Item 4: Intensive education for low salt diet induces the significant decrease of blood pressure in Intervention group compared to control group.
4. Study Flow

   * Period

     1. Washout period (-8 weeks;Point 0 to 0 weeks; Point 1)
     2. Olmesartan Period ( 0 week; point 1 to 8 weeks; point 2)
     3. Intervention period (8 week ; point 2 to 16 weeks; point 3)
   * For patients with taking ACEI, other ARB, diuretics, or renin inhibitor, already; Initial wash-out period for 8 weeks, and then (point 1) prescription of Olmesartan 40 mg qd for 8 weeks, and then (point 2) allocation to Intensive group or control group for 8 weeks, and then the study will be over (point 3).
   * For patients without taking ACEI, other ARB, diuretics, or renin inhibitor; For initial 8 weeks, adjust the blood pressures around 140/90 mmHg, and then (point 1) prescription of Olmesartan 40 mg qd for 8 weeks, and then (point 2) allocation to Intensive group or control group for 8 weeks, and then the study will be over (point 3).
   * Blood pressure control Adjust the blood pressures around 140/90 mmHg with other hypertensive drugs except ACEI, other ARB, diuretics, or renin inhibitor during whole period.
   * Intensive diet education:

For 8 weeks, dietitian will call patients to take the information according to pre-defined questionnaire, to check the daily diet habit and daily food taken, and to guide how to lessen sodium intake for 30 min at each call. The call will be done once a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19 years or more and 75 years or less
* Hypertension patients: Patients whose blood pressure is 140/90mmHg and over, patients is newly diagnosed with hypertension or is prescribed antihypertensive medications.
* Hypertensive patients verified 2 times or more of albuminuria 30 mg/g cr or more in a spot urine sample with interval of 1 week or more in recent 6 months
* Estimated glomerular filtration rate (GFR) by Modification of Diet in Renal Disease (MDRD) equation 30 ml/min/1.73 m2 or more
* Patients who give written consent to this study by oneself

Exclusion Criteria:

* Blood pressure more than 160/100 mmHg
* Pregnant
* Serum potassium level more than 5.5 mEq/L at screening period
* Patients with malignancy, acute cerebral infarction, acute myocardial infarction, unstable angina, percutaneous coronary arterial intervention (PCI), or coronary artery bypass graft (CABG) in recent 6 months
* Patients with diabetes mellitus
* Patients who have an allergy to Olmesartan
* Patients who were involved in other clinical trial in recent 1 month or are participated in screening period
* Patients taking medication(s) of corticosteroid or immunosuppressant in a screening period

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ho Jun Chin, PhD, Principal Investigator — Seoul National University Bundang Hospital; Chun-Soo Lim, PhD, Study Chair — SMG-SNU Boramae Medical Center; Dong Ki Kim, PhD, Principal Investigator — Seoul National University Hospital; Suhnggwon Kim, PhD, Principal Investigator — Seoul National University Hospital; Bum Soon Choi, PhD, Principal Investigator — Seoul St. Mary's Hospital; Sang-Ho Lee, PhD, Principal Investigator — Kyunghee University; Jung-Hwan Park, PhD, Principal Investigator — Konkuk University; Sung Joon Shin, PhD, Principal Investigator — DongGuk University
Locations (7):
- South Korea (7):
  - Seoul National University Bundang Hospital, Seongnam, Kyeong Ki
  - Dongguk University Ilsan Hospital, Ilsan, Kyeongki
  - Seoul National University Hospital, Seoul, Seoul
  - Kyung Hee University, Seoul, Seoul
  - Seoul St. Mary's Hospital, Seoul, Seoul
  - Konkuk University School of Medicine, Seoul, Seoul
  - SMG-SNU Boramae Medical Center, Seoul, Seoul

REFERENCES:
- [Background] Vogt L, Waanders F, Boomsma F, de Zeeuw D, Navis G. Effects of dietary sodium and hydrochlorothiazide on the antiproteinuric efficacy of losartan. J Am Soc Nephrol. 2008 May;19(5):999-1007. doi: 10.1681/ASN.2007060693. Epub 2008 Feb 13. PMID 18272844
- [Background] Ekinci EI, Thomas G, Thomas D, Johnson C, Macisaac RJ, Houlihan CA, Finch S, Panagiotopoulos S, O'Callaghan C, Jerums G. Effects of salt supplementation on the albuminuric response to telmisartan with or without hydrochlorothiazide therapy in hypertensive patients with type 2 diabetes are modulated by habitual dietary salt intake. Diabetes Care. 2009 Aug;32(8):1398-403. doi: 10.2337/dc08-2297. Epub 2009 Jun 23. PMID 19549737
- [Background] He FJ, Marciniak M, Visagie E, Markandu ND, Anand V, Dalton RN, MacGregor GA. Effect of modest salt reduction on blood pressure, urinary albumin, and pulse wave velocity in white, black, and Asian mild hypertensives. Hypertension. 2009 Sep;54(3):482-8. doi: 10.1161/HYPERTENSIONAHA.109.133223. Epub 2009 Jul 20. PMID 19620514
- [Background] Intersalt: an international study of electrolyte excretion and blood pressure. Results for 24 hour urinary sodium and potassium excretion. Intersalt Cooperative Research Group. BMJ. 1988 Jul 30;297(6644):319-28. doi: 10.1136/bmj.297.6644.319. PMID 3416162
- [Background] Swift PA, Markandu ND, Sagnella GA, He FJ, MacGregor GA. Modest salt reduction reduces blood pressure and urine protein excretion in black hypertensives: a randomized control trial. Hypertension. 2005 Aug;46(2):308-12. doi: 10.1161/01.HYP.0000172662.12480.7f. Epub 2005 Jun 27. PMID 15983240
- [Derived] Hwang JH, Oh S, Chin HJ, Kim S, Kim DK, Kim S, Park JH, Shin SJ, Lee SH, Choi BS, Lim CS. Comparison of the performance of currently used estimated glomerular filtration rate equations with 24-hour urine creatinine clearance: sample analysis of randomised controlled trial participants. BMJ Open. 2023 Aug 23;13(8):e067398. doi: 10.1136/bmjopen-2022-067398. PMID 37612109
- [Derived] McMahon EJ, Campbell KL, Bauer JD, Mudge DW, Kelly JT. Altered dietary salt intake for people with chronic kidney disease. Cochrane Database Syst Rev. 2021 Jun 24;6(6):CD010070. doi: 10.1002/14651858.CD010070.pub3. PMID 34164803
- [Derived] Conley MM, McFarlane CM, Johnson DW, Kelly JT, Campbell KL, MacLaughlin HL. Interventions for weight loss in people with chronic kidney disease who are overweight or obese. Cochrane Database Syst Rev. 2021 Mar 30;3(3):CD013119. doi: 10.1002/14651858.CD013119.pub2. PMID 33782940
- [Derived] An JN, Hwang JH, Lee JP, Chin HJ, Kim S, Kim DK, Kim S, Park JH, Shin SJ, Lee SH, Choi BS, Lim CS. The Decrement of Hemoglobin Concentration with Angiotensin II Receptor Blocker Treatment Is Correlated with the Reduction of Albuminuria in Non-Diabetic Hypertensive Patients: Post-Hoc Analysis of ESPECIAL Trial. PLoS One. 2015 Jun 22;10(6):e0128632. doi: 10.1371/journal.pone.0128632. eCollection 2015. PMID 26098847
- [Derived] Baek SH, Kim S, Kim DK, Park JH, Shin SJ, Lee SH, Choi BS, Chin HJ, Kim S, Lim CS. A low-salt diet increases the estimated net endogenous acid production in nondiabetic chronic kidney disease patients treated with angiotensin receptor blockade. Nephron Clin Pract. 2014;128(3-4):407-13. doi: 10.1159/000369558. Epub 2014 Dec 18. PMID 25531146

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were selected from 7 centers in Korea (Seoul National University Boramae Medical Center, Seoul National University Bundang Hospital, Seoul National University Hospital, Konkuk University Hospital, Dongguk University Ilsan Hospital, Kyung Hee University Medical Center, and Seoul St. Mary's Hospital) and enrolled from Mar. 2012 to Mar. 2013.
Pre-assignment Details: We screened 312 patients before 8 weeks of study initiation, and 269 patients were enrolled. During the 1st 8 weeks of this study (ARB run-in), 13 patients were withdrawn. After that, 256 patients were randomized, 11 participants were dropped out between 8th week and 16th week, and 245 who completed the trial were included in the analysis .
Groups:
- Conventional Education of Low-salt Diet Group: Education for low salt diet will be conducted as in office with brief communication with a patient and a physician.
- Intensive Education of Low-salt Diet Group: For 8 weeks, dietitian will call patients to take the information according to pre-defined questionnaire, to check the daily diet habit and daily food taken, and to guide how to lessen sodium intake for 30 min at each call. The call will be done once a week for 8 weeks.
  Intensive education for low salt diet : For 8 weeks, dietitian will call patients to take the information according to pre-defined questionnaire, to check the daily diet habit and daily food taken, and to guide how to lessen sodium intake for 30 min at each call. The call will be done once a week for 8 weeks.
Period: Overall Study
Arm/Group | Conventional Education of Low-salt Diet Group | Intensive Education of Low-salt Diet Group
Started | 131 (A total of 13 patients were withdrawn from 269 patients. The remained 256 patients were randomized.) | 125
Completed | 126 | 119
Not Completed | 5 | 6
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — diagnosed DM | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Education of Low-salt Diet Group | Intensive Education of Low-salt Diet Group | Total
Number analyzed (Participants) | 131 | 125 | 256
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 107 | 116 | 223
  >=65 years | 24 | 9 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (14.3) | 48.2 (12.2) | 49.5 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 54 | 118
  Male | 67 | 71 | 138
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 131 | 125 | 256

OUTCOME MEASURES:

1. Primary Outcome: ∆Albuminuria by 24-hour Urine Protein Excretion
Description: Change in albuminuria as a 24-hour urine protein excretion by intensive education of low salt diet during taking olmesartan
  *In outcome measure data table, the 24-hour urine collection at 16th week was omitted in 3 out of 245 patients (1 for intensive education group and 2 for conventional education group). Values of each study week were "mean" of all participants on specific study week, but "∆albuminuria (week 8 - week 16)" value was "mean" of ∆ values of "8 weeks-16 weeks" in each individuals. Therefore, values of 3 patients were excluded in "mean of ∆albuminuria (week 8 - week 16)". That's why simple subtraction (week 8 - week 16) of values are not matched with the data.
Time Frame: changes from week 8 at week 16 (week 8 - week 16)
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Conventional Education of Low-salt Diet Group | Intensive Education of Low-salt Diet Group
Number analyzed (Participants) | 126 | 119
mg/day
  24hr-urine albumin (8th week) | 483.5 (646.7) | 569.9 (718.9)
  24hr-urine albumin (16th week);n=124, 118 | 487.3 (688.8) | 417.4 (597.0)
  Mean of ∆albuminuria (week 8-week 16); n=124, 118 | -0.4 (371.9) | 154.0 (489.6)
Statistical Analysis 1: Comparison: Conventional Education of Low-salt Diet Group vs Intensive Education of Low-salt Diet Group; Differences with two-tailed P<0.05 were considered statistically significant; Test type: Superiority or Other; p = 0.006, t-test, 2 sided — for albuminuria changes from week 8 at week 16 (week 8 - week 16)
Statistical Analysis 2: Comparison: Conventional Education of Low-salt Diet Group; Test type: Superiority or Other; p = 0.99, Mixed Models Analysis — for 24-hour urine albumin excretion between 8 weeks and 16 weeks
Statistical Analysis 3: Comparison: Intensive Education of Low-salt Diet Group; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — for 24-hour urine albumin excretion between 8 weeks and 16 weeks in intensive education group

2. Secondary Outcome: ∆Hemoglobin (0 Week - 16 Weeks)
Description: The change of hemoglobin after prescription of Olmesartan
Time Frame: 0 week, 16 weeks
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Conventional Education of Low-salt Diet Group | Intensive Education of Low-salt Diet Group
Number analyzed (Participants) | 126 | 119
g/dL
  Hemoglobin (week 0) | 13.8 (1.7) | 14.0 (1.8)
  Hemoglobin (week 8) | 13.5 (1.8) | 13.7 (1.7)
  Hemoglobin (week 16) | 13.3 (1.7) | 13.4 (1.7)
  Hemoglobin changes from week 0 at week 16 | 0.46 (0.90) | 0.62 (0.96)
Statistical Analysis 1: Comparison: Conventional Education of Low-salt Diet Group vs Intensive Education of Low-salt Diet Group; Test type: Superiority or Other; p = 0.187, t-test, 2 sided — for hemoglobin changes from week 0 at week 16 (week 0 - week 16)

3. Secondary Outcome: Na Excretion Change in 24 Hour-urine Collection Between Weeks 8 and 16
Description: Change of sodium excretion rate in 24 hour-urine collection by intensive education for low salt diet at week 16
Time Frame: week 8 and week 16
Measure: Mean (Standard Deviation); unit: mEq/day
Arm/Group | Conventional Education of Low-salt Diet Group | Intensive Education of Low-salt Diet Group
Number analyzed (Participants) | 126 | 119
mEq/day
  week 8 | 155.5 (71.1) | 157.4 (74.7)
  week 16; n=124, 118 | 147.1 (66.1) | 122.1 (59.9)
  ∆Na excretion (week 8 - week 16);n=124, 118 | 9.0 (54.5) | 35.4 (64.4)
Statistical Analysis 1: Comparison: Conventional Education of Low-salt Diet Group vs Intensive Education of Low-salt Diet Group; Test type: Superiority or Other; p = 0.001, t-test, 2 sided — for changes from week 8 at week 16 (week 8 - week 16)

4. Secondary Outcome: Systolic and Diastolic Blood Pressure Change Between Weeks 8 and 16
Description: Change in Systolic and Diastolic Blood Pressure from Week 8 to Week 16 in the Intensive Education Group compared to the Conventional Education Group
Time Frame: week 8 and week 16
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Conventional Education of Low-salt Diet Group | Intensive Education of Low-salt Diet Group
Number analyzed (Participants) | 126 | 119
mm Hg
  Systolic BP at week 8 | 121.8 (18.4) | 122.1 (14.0)
  Systolic BP at week 16 | 121.2 (14.9) | 120.4 (14.9)
  sBP changes from week 8 at week 16 | 0.6 (15.1) | 1.7 (14.6)
  Diastolic BP at week 8 | 73.4 (11.6) | 73.6 (11.0)
  Diastolic BP at week 16 | 74.8 (10.5) | 73.1 (10.4)
  dBP changes from week 8 at week 16 | -0.7 (10.0) | 0.5 (9.8)
Statistical Analysis 1: Comparison: Conventional Education of Low-salt Diet Group vs Intensive Education of Low-salt Diet Group; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — for sBP changes from week 8 at week 16 (week 8 - week 16)
Statistical Analysis 2: Comparison: Conventional Education of Low-salt Diet Group vs Intensive Education of Low-salt Diet Group; Test type: Superiority or Other; p = 0.585, t-test, 2 sided — for dBP changes from week 8 at week 16 (week 8 - week 16)

ADVERSE EVENTS:
Time Frame: from week 8 to week 16 (for 8 weeks)
Arm/Group | Conventional Education of Low-salt Diet Group | Intensive Education of Low-salt Diet Group
Serious Adverse Events (participants affected / at risk) | 0/131 | 0/125
Other Adverse Events (participants affected / at risk) | 1/131 | 2/125
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Education of Low-salt Diet Group (N=131) | Intensive Education of Low-salt Diet Group (N=125)
Elevated serum creatinine (Renal and urinary disorders) | 0 (0) | 2 (2) — Elevation of serum creatinine level : Physician assessed ARB could not be continued
Headache (Nervous system disorders) | 1 (1) | 0 (0) — Headache

LIMITATIONS AND CAVEATS:
The major limitation of this study is that we used a 24-hour volume urine collected at a single time point for each follow-up visit. Urine excretion can be influenced by the sodium intake of individual patients at certain point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No